CLINICAL TRIAL: NCT01994122
Title: Mental Health and Resilience in Emerging Adulthood
Status: Terminated | Type: Observational
Why Stopped: The study has been terminated because of recruitment difficulties and lack of further funding
Sponsor: University of Tromso (Other)
Collaborators: Harstad University College (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013/101(REK)
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Depression; Anxiety; Personality Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Personality Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- People who have dropped out of school
- College students (control group)

SUMMARY:
The purpose of this study is to examine differences in selected psychiatric/psychological variables between a sample of unemployed young adults who have dropped out of high school and a sample of college students.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-25 years old who have dropped out of school and who are currently unemployed

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects 18-25 years old who have dropped out of school and who are currently unemployed
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of axis-1 disorders in the sample. | Within 6 months of enrolment
  Participants will be subject to an assessment with the MINI International Neuropsychiatric Interview, resulting in an overview of axis-1 psychiatric disorders in the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Wynn, ph.d., Principal Investigator — University of Tromsø, Norway
Locations (1):
- Harstad University Colle, Harstad, Norway